CLINICAL TRIAL: NCT05056545
Title: Implementation and Evaluation of a Large-scale Postpartum Family Planning Program in Rwanda
Brief Title: Postpartum Family Planning Program in Rwanda
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kristin Wall, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002354; R01HD101600 (NIH)
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Family Planning
Keywords: Postpartum; Intrauterine Device; Long-acting reversible contraception

STUDY DESIGN:
Intervention Model Description: This step-wedge clinical trial will train all nurse/midwives working in antenatal care (ANC), labor and delivery (L&D), infant vaccination (IV), or postpartum services at one of the study facilities in PPFP promotions or provision. The study team will train 'Happy Clients' (postpartum women who received promotions and selected a PPFP method) and community health workers affiliated with the intervention facilities as PPFP promotional agents. Women eligible for PPFP services in this study will be at any stage of pregnancy or up to 14 weeks postpartum, and receiving ANC, L&D, IV, or postpartum services at one of the intervention facilities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPFP Intervention (Experimental): The study team will train government clinic staff in ANC, L&D, IV, or postpartum services to promote and provide the PPFP intervention at the selected facilities. Community Health Workers (CHW) and 'Happy Clients' will be trained as PPFP promotional agents. Video-based PPFP promotions will be shown at the intervention facilities. If interested in PPFP, women will be referred to the facility by their CHW.
  Interventions: Behavioral: C4 Intervention
- Standard of Care (No Intervention): Currently, no systematic PPFP training, promotional, or service delivery activities are regularly taking place at the selected facilities. The team will compare the intervention with historical records from the facilities applying intervention and compare

INTERVENTIONS:
Behavioral: C4 Intervention — C4 Intervention, is an innovative form of Post Partum Family Planning (PPFP). PPFP methods include: the copper intrauterine device, hormonal implant, tubal ligation, and (after 6 weeks post-partum in breastfeeding women) Depo-Provera and oral contraceptive pills. These are provided as current, standard of care in Rwanda, are procured by the government, and administered by trained nurses and doctors.
  The C4 training will occur at the 4 pilot facilities. Training will include a 2-day didactic session covering PPFP provision, follow-up, use of the C4 counseling flipchart; mock counseling sessions; and PPIUD and PP implant insertion and removal trainings. The study team will train government clinic staff in family planning, ANC, L&D, and IV to promote C4 at the selected facilities. 'Happy Clients' will be recruited from women who received promotions and selected PPFP to join a clinic-based PPFP promotions team. Women interested in PPFP will be referred to the facility by their CHW.
  Arms: PPFP Intervention

SUMMARY:
This trial wants to address high unmet need for postpartum family planning (PPFP) in Rwanda. A previous pilot study tested the intervention (informed by formative work with couples/clients, clinic providers, champions, and community health workers), which significantly increased the use of PPFP in government clinics. This study now proposes to use an implementation science framework to test the hypothesis that the proposed PPFP intervention is adaptable to large-scale implementation, cost-effective, and sustainable. This PPFP could dramatically reduce unintended pregnancy and abortion and improve birth spacing and maternal and newborn health.

DETAILED DESCRIPTION:
In 2017-2018, the study team worked closely with the Rwanda Ministry of Health (MOH) to develop and pilot test a theory-based, multi-level intervention targeting postpartum family planning (PPFP) supply and demand in 4 government health facilities in Kigali, the capital. This innovative PPFP intervention was informed by clients, clinic providers, champions, and Community Health Workers. Long-acting reversible contraceptives (LARC), the intrauterine device (PPIUD) and implant, are fundamental to PPFP programs. LARCs are highly effective and are the only reversible methods that may be safely used in early postpartum period by breastfeeding women. During the pilot, LARC uptake among postpartum women increased significantly (172% for PP implant, 2,687% for PPIUD), PPFP feasibility and acceptability were high among providers and clients, and side-effects were rare.

The study team now proposes to use an implementation science framework to evaluate the effectiveness of different PPFP demand creation strategies and test the hypothesis that our PPFP intervention is adaptable to large-scale implementation, cost-effective, and sustainable. In a Type 2 effectiveness-implementation hybrid study, we will evaluate facility organizational readiness prior to implementing the PPFP intervention in a clinic randomized trial in 10 high-volume health facilities in Kigali, Rwanda (Aim 1). Adaptability and sustainability within government facilities is a critical aspect of the proposal, and the MOH and other local stakeholders will be engaged from the outset. It is expected that this project will deliver PPFP counseling to over 21,000 women/couples during the project period. They will then evaluate the PPFP intervention effectiveness and implementation processes using RE-AIM (Aim 2). The team hypothesizes that the PPFP intervention will significantly increase the number of stakeholders engaged, PPFP providers and promoters, couples/clients receiving information about PPFP (reach), and LARC uptake (effectiveness) comparing intervention versus standard of care. It is expected that PPFP client satisfaction will be high and side-effects will be rare. The independent effectiveness of each demand creation strategy on LARC uptake will be estimated. Assessment of measures of PPFP intervention adoption, implementation, and maintenance at the patient-, provider- and stakeholder-level to assess PPFP intervention sustainability will be completed by the study team. Finally, this project will evaluate PPFP intervention cost-effectiveness and develop a national costed implementation plan to guide Rwandan MOH decision-making for nationwide roll-out of PPFP services (Aim 3). This trial hypothesizes that the PPFP intervention will be cost-saving relative to standard of care.

This intervention represents an important contribution to the Rwanda Family Planning 2020 goals and the MOH are enthusiastic to see our successful pilot efforts expanded to a larger number of facilities for greater and sustained impact. The new PPFP implementation model is designed to be replicable and expandable to other countries in the region which similarly have high unmet need for PPFP.

ELIGIBILITY:
Inclusion Criteria:

* Eligible PPFP promoters will be government facility providers working in ANC,L&D, IV and/or postpartum services at one of the study facilities.
* Eligible PPFP providers will be government facility providers working in L&D, and/or family planning services at one of the study facilities.
* Eligible Happy Client promotors will be postpartum women who received promotions and selected a PPFP method.
* Eligible nurse/midwife and CHW promotors will be women working as nurses or CHWs at one of the intervention facilities.
* All women eligible for PPFP services in this study will be at any stage of pregnancy or up to 14 weeks postpartum, and receiving antenatal care (ANC), L&D, IV, or postpartum services at one of the intervention or pilot facilities

Exclusion Criteria:

* Prisoners

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26215 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Numbers of clinic directors engaged | Through study completion, an average of 3 years
  Numbers of clinic directors engaged to provide the PPFP Intervention
Number of Nurses trained to promote PPFP | After completion of a 2-day training
  The number of nurses who complete PPFP intervention session to promote PPFP use
Number of CHWs trained to promote PPFP | After completion of a 2-day training session
  The number of CHWs who complete C4 training session to promote PPFP use
Number of providers trained to provide PPFP | After completion of a 2-day training session
  Nurses and midwives working labor and delivery and family planning will attend a 2-day didactic training session. Providers will complete a post-training test consisting of 10 true or false questions. Those who do not score at least 80% on the post-training test will be offered re-training after one week.
Number of providers certified to provide PPFP | After completion of a 2-day training session
  After completing the didactic training, providers will have the opportunity to become certified, by correctly inserting 5 PPIUDs and 5 PP implants under supervision.
Number of promotions to pregnant or postpartum women/couples | Beginning at the first antenatal care visit up to post-partum week 14 (up to 54 weeks)
  The number of pregnant or postpartum women/couples receiving one-on-one C4 counseling
Number of PPIUD insertions | Up to postpartum week 14
  The number of postpartum women who opt to have a PPIUD inserted
Number of PP implant insertions | Up to postpartum week 14
  The number of postpartum women who opt to have a PP implant inserted.

SECONDARY OUTCOMES:
Cost-effectiveness/cost-utility: Couple Years Protection (CYP) | Years 2 and 4 of the project period
  Cost, in US dollars adjusted for the year of data analysis per CYP
Cost-effectiveness/cost-utility: Cost per Quality Adjusted life years (QALY) | Years 2 and 4 of the project period
  Cost, in US dollars adjusted for the year of data analysis of cost per QALY saved

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Wall, PhD, Principal Investigator — Emory University
Locations (1):
- Project San Francisco, Kigali, Kigali, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification
Supporting Information: Study Protocol
Time Frame: Immediately following publication, ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal and whose proposed use of the data has been approved by the Rwanda National Ethics Committee, to achieve the aims in the approved proposal. Proposals should be directed to kmwall@emory.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Wall KM, Ingabire R, Mazzei A, Umuhoza C, Parker R, Tichacek A, Nizam A, Sales JM, Haddad LB, Corso P, Allen S, Nyombayire J, Karita E. Implementation and evaluation of a large-scale postpartum family planning program in Rwanda: study protocol for a clinic-randomized controlled trial. Trials. 2022 Apr 22;23(1):337. doi: 10.1186/s13063-022-06261-5. PMID 35459259